CLINICAL TRIAL: NCT05261841
Title: Observational Analysis and Elaboration of a Predictive Model on the Effects of Physical Activity and Individual Lifestyles in the Management of Diabetic Disease Type 2 as Part of the GATEKEEPER H2020 Project.
Brief Title: Predictive Model on the Effect of Lifestyles in the Management of T2D
Acronym: GK_T2D
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Casa Sollievo della Sofferenza IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: GATEKEEPER-V1.6_03 DIC 2020
Record Dates: First submitted 2022-02-15; First posted 2022-03-02 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Type 2 Diabetes
Keywords: T2D; CONSUMER DEVICES; SMARTWATCH; ARTIFICIAL INTELLIGENCE
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TYPE 2 DIABETES: Patients affected by type 2 diabetes
  Interventions: Other: Standard care for T2D patients, Smartwatch

INTERVENTIONS:
Other: Standard care for T2D patients, Smartwatch — No intervention, observational study

SUMMARY:
This study aims to produce new evidence on the positive effects of physical activity and certain individual lifestyles in the control of type 2 diabetic disease. The goal is to build and evaluate the effectiveness of a new parsimonious risk prediction model based on the use of classical variables (blood exams), already used in other models for predicting the risk related to the disease, together with measures obtained from the use of wearable devices (steps count, sleep hours, heart rate).

DETAILED DESCRIPTION:
Scientific literature has shown that the use of wearable devices can improve the control of type 2 diabetes mellitus. The aim of the study is to develop a statistical model for the control of type 2 diabetes mellitus (DMT2) based on the use of "conventional" clinical parameters and the use of "unconventional" data from wearable devices. The medical outcome variable that will be used to measure diabetes control and model performance will be the Glycated Hemoglobin (HbA1c). The participant will receive a Samsung smartwatch (Galaxy Watch 3) and a Samsung smartphone (A51), (the latter only in case the participant is not in possession of a compatible smartphone) which he/she must wear during his daily activities and also during the night to measure daily activity, sleep hours and heart rate. Casa Sollievo della Sofferenza Hospital previoulsy developted the ENFORCE calculator, an inexpensive and parsimonious prediction model of 2-year all cause mortality in real life patients with T2D. In this study the investigators aim to elaborate a standardized validated risk scores similar to what has been done for ENFORCE.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 55 years old
* Affected by Type 2 Diabetes and monitored by Casa Sollievo della Sofferenza Hospital
* Basic skills in using a smartphone and its apps
* Available to use the device and its applications
* Ability to understand the informed consent

Exclusion Criteria:

* Inability to understand the informed consent
* Low life expectancy
* Type 1 Diabetes
* Secondary Diabetes

Ages: 55 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes followed by Casa Sollievo della Sofferenza Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-06-26 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline HbA1c at 6 and 12 months | Baseline, 6 months, 12 months
  Glycated Hemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore De Cosmo, MD, Principal Investigator — Casa Sollievo della Sofferenza IRCCS
Locations (1):
- Casa Sollievo della Sofferenza IRCCS, San Giovanni Rotondo, FG, Italy

REFERENCES:
- [Background] Copetti M, Shah H, Fontana A, Scarale MG, Menzaghi C, De Cosmo S, Garofolo M, Sorrentino MR, Lamacchia O, Penno G, Doria A, Trischitta V. Estimation of Mortality Risk in Type 2 Diabetic Patients (ENFORCE): An Inexpensive and Parsimonious Prediction Model. J Clin Endocrinol Metab. 2019 Oct 1;104(10):4900-4908. doi: 10.1210/jc.2019-00215. PMID 31087060
- See also: This study is currently in the frame of Horizon2020 GATEKEEPER project, that is a European Multi Centric Large-Scale Pilot on Smart Living Environments. — http://www.gatekeeper-project.eu/